CLINICAL TRIAL: NCT01199848
Title: Effect of Strawberry on Oxidative Stress- and Inflammatory-mediated Insulin Resistance (IR) in Humans: Combating a Major Risk Factor for Diabetes and Cardiovascular Disease Through Diet
Brief Title: A Study of Strawberries and Disease Risk
Acronym: STRB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: California Strawberry Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STRB 2010-033
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Nutritional and Metabolic Diseases; Inflammation; Physiological Responses
Keywords: nutrition; polyphenolic; strawberry; insulin resistance; metabolic syndrome
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Inflammation; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Pbo
  Interventions: Dietary Supplement: Placebo
- 10G STRB powder (Experimental): Dose 1
  Interventions: Dietary Supplement: 10G
- 20G STRB powder (Experimental): Dose 2
  Interventions: Dietary Supplement: 20G
- 40G STRB powder (Experimental): Dose 3
  Interventions: Dietary Supplement: 40G
- PlacebonoFiber (Placebo Comparator): Placebo without fiber
  Interventions: Dietary Supplement: Placebonofiber

INTERVENTIONS:
Dietary Supplement: Placebo — whole milk shake without strawberry powder served with the high fat/carbohydrate test meal
  Other Names: Pbo
  Arms: Placebo
Dietary Supplement: 10G — whole milk shake with 10g strawberry powder served with the high fat/carbohydrate test meal
  Other Names: Dose 1
  Arms: 10G STRB powder
Dietary Supplement: 20G — whole milk shake with 20 strawberry powder served with the high fat/carbohydrate test meal
  Other Names: Dose 2
  Arms: 20G STRB powder
Dietary Supplement: 40G — whole milk shake with 40g strawberry powder served with the high fat/carbohydrate test meal
  Other Names: Dose 3
  Arms: 40G STRB powder
Dietary Supplement: Placebonofiber — Placebo without Fiber
  Arms: PlacebonoFiber

SUMMARY:
The purpose of this study is to test whether compounds found in strawberries (polyphenolics which are typically found in berry products, tea, coffee, red wine, and chocolate) will help reduce insulin resistance and inflammation, known factors in your blood associated with disease risk, when eaten with a standard high fat/carbohydrate meal.

DETAILED DESCRIPTION:
The main study is a single-center, randomized, cross-over, 4-arm, dose-response, single- blinded, 6-hour postprandial study to evaluate the ability of strawberry powder to block meal-induced oxidative stress and inflammation and concomitantly improve postprandial insulin sensitivity and glucose handling.

A planned sample size of 45 will be recruited into the study. Thirty subjects for the main study and 15 subjects for the complement study. Subjects can participate in both studies and if subjects participate in both studies, there will be a time gap between the main study and the complement study due to the volume of blood permitted to collect within 56 days.

The complement study will be a 2-arm placebo controlled study following the exact same protocol as the main study, but using only one strawberry dose (Dose 3 as in the main study) and comparing the effects relative to a placebo that does not control for fiber.

The main study will take 5- 6 weeks per subject to complete and the complement study will take 1-2 weeks per subject to complete, depending on subject's schedule.

The procedures conducted at the screening visit include blood sampling by finger prick for a fasting blood sugar test and anthropometric measurements (height, weight, and waist circumference), vital sign measurements (blood pressure and heart rate) and completion of a series of questionnaires relating to volunteers' general health and eating habits. Volunteers may be asked to complete an oral glucose/sugar tolerance test (OGTT) at screening. Volunteers will be exempt from the OGTT procedure if other qualifying conditions are present. Briefly, subjects undergoing OGTT will be asked to drink a glucose drink (similar in taste to kool-aid) in the morning after a 10 hour fast. Blood glucose finger pricks will then be done at 1 hour and 2 hours for determination of glucose tolerance. If the OGTT is necessary, additional compensation will be provided.

If qualified, subjects will undergo a 7-day pre-study period during which they will be asked to record their usual diet intake for 3 days, including 2 weekdays and 1 weekend day, EITHER followed by randomization into 1 of 4 treatment beverage sequences for the main study: Placebo (Pbo), Strawberry Dose 1, Strawberry Dose 2 and Strawberry Dose 3, OR followed by randomization into 1 of 2 treatment (Placebo without fiber and Strawberry Dose 3) beverage sequences for the complement study.

We expect it to be very difficult to eliminate or severely restrict polyphenolic diet during the entire study period, therefore subjects will be asked to limit only berry product intake during the study period. However, subjects will be asked to limit all polyphenolic foods in their diet for 3 days prior to each study visit.

All subjects will consume the standard high fat/ carbohydrate meal (known to induce oxidative- and inflammatory- stress) accompanied by 1 of 4 test beverages (whole milk shake with or without strawberry powder) on four separate occasions for the main study OR 1 of 2 test beverages on two separate occasions for the complement study, so that each subject will serve as their own control.

Subjects will arrive at the study visits fasted for at least 10 hours, well hydrated and rested. Each study visit will require blood draws throughout the visit. After pre-study procedures (height, weight, waist circumference, blood pressure, blood glucose finger prick) and while fasting, a registered nurse (RN) will place a catheter (flexible tubing) in subjects' arm for the purpose of drawing blood. This catheter will remain only throughout the study day. Approximately 1 tablespoon of blood will be taken at this time. The test meal and strawberry shake will be served and thereafter subjects will have blood draws (1 T each time) at designated time points for the next 6 hours. Each visit will last approximately 7 hours and subjects will be required to remain at the Clinical Nutrition Research Center on the IIT Campus for the duration of the visit. Blood samples will be collected at designated time points during the postprandial period for analysis of metabolic (insulin and glucose homeostasis), oxidative and inflammatory endpoint markers.

ELIGIBILITY:
Inclusion Criteria:

Eligible volunteers must meet ONE or MORE of the criteria (numbers 1-4) associated with insulin resistance along with all of the other criteria listed (numbers 5-9):

1. Blood glucose concentration between140-199 mg/dL at 2hr from OGTT.
2. Elevated fasting glucose (≥110 mg/dL and <126 mg/dL)
3. Elevated fasting insulin (>75th percentile cutoff of 13.13 μU/mL)
4. Insulin resistance defined by the homeostasis model assessment method of insulin resistance (HOMA-IR) (glucose [in millimoles per liter] × insulin [in microunits per milliliter]/22.5) values of at least 2.5.
5. Waist circumference >102 cm (men) and > 88 cm (women) for screening visit invitation because many epidemiology studies have been shown that waist circumferences may be related to insulin resistance.
6. Nonsmokers
7. Not taking any medications that would interfere with outcomes of the study, i.e. lipid lowering medications, anti-inflammatory drugs, or dietary supplements
8. 18 years of age and older
9. No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease

Exclusion Criteria:

* Pregnant and/or lactating
* Allergy or intolerance to strawberries and dairy products.
* Current regular consumption of strawberries is > 2 servings per day.
* Fasting blood glucose ≥ 126 mg/dL. Subjects identified with elevated fasting blood glucose levels will be advised to contact their primary care physician for appropriate follow-up care.
* Taking over the counter antioxidant supplements or other supplements that may interfere with the study procedures or endpoints.
* Subjects with unusual dietary habits (e.g. pica).
* Actively losing weight or trying to lose weight (unstable body weight fluctuations of > 5 kg in a 60 day period).
* Excessive exercisers or trained athletes.
* Subjects with documented atherosclerotic disease, inflammatory disease, diabetes mellitus, or other systemic diseases.
* Addicted to drugs and/or alcohol.
* Medically documented psychiatric or neurological disturbances.
* Smoker (past smoker may be allowed if cessation is > 2 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2015-10-15 (Actual); Study Completion 2015-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indika Edirisinghe, PhD, Principal Investigator — Institute for Food Safety and Health; Britt Burton-Freeman, PhD, MS, Principal Investigator — Institute for Food Safety and Health
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton-Freeman B, Linares A, Hyson D, Kappagoda T. Strawberry modulates LDL oxidation and postprandial lipemia in response to high-fat meal in overweight hyperlipidemic men and women. J Am Coll Nutr. 2010 Feb;29(1):46-54. doi: 10.1080/07315724.2010.10719816. PMID 20595645
- [Derived] Park E, Edirisinghe I, Wei H, Vijayakumar LP, Banaszewski K, Cappozzo JC, Burton-Freeman B. A dose-response evaluation of freeze-dried strawberries independent of fiber content on metabolic indices in abdominally obese individuals with insulin resistance in a randomized, single-blinded, diet-controlled crossover trial. Mol Nutr Food Res. 2016 May;60(5):1099-109. doi: 10.1002/mnfr.201500845. Epub 2016 Mar 29. PMID 26842771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Chicago, IL, USA from September 2010 to January 2013.
Pre-assignment Details: 7-day pre-study period: Following the screening visit, qualified subjects were asked to record their usual diet intake for 3 days, including 2 weekdays and 1 weekend day in order to know their usual intake and to coach them on what foods in their diet are rich in polyphenolics, especially 3 days prior to their each study visit.
Groups:
- All Study Participants: All participants received all 4 interventions (Placebo, STRB 10g, STRB 20g, and STRB 40g) in a randomized sequence
  Placebo: whole milk shake without strawberry powder served with the high fat/carbohydrate test meal Dose 1-10G: whole milk shake with 10g strawberry powder served with the high fat/carbohydrate test meal Dose 2- 20G: whole milk shake with 20 strawberry powder served with the high fat/carbohydrate test meal Dose 3-40G: whole milk shake with 40g strawberry powder served with the high fat/carbohydrate test meal
Period: Placebo Arm
Arm/Group | All Study Participants
Started | 29
Completed | 21
Not Completed | 8
Period: 10g STR Arm
Arm/Group | All Study Participants
Started | 21
Completed | 21
Not Completed | 0
Period: 20G STRB Arm
Arm/Group | All Study Participants
Started | 21
Completed | 21
Not Completed | 0
Period: 40G STRB Arm
Arm/Group | All Study Participants
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subject characteristics were analyzed using descriptive statistics and tabulated.
Groups:
- All Participants: All participants received all 4 interventions (Placebo, STRB 10g, STRB 20g, and STRB 40g) in a randomized sequence Placebo: whole milk shake without strawberry powder served with the high fat/carbohydrate test meal Dose 1-10G: whole milk shake with 10g strawberry powder served with the high fat/carbohydrate test meal Dose 2- 20G: whole milk shake with 20 strawberry powder served with the high fat/carbohydrate test meal Dose 3-40G: whole milk shake with 40g strawberry powder served with the high fat/carbohydrate test meal
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Insulin Levels for 6 Hours
Description: Strawberry dose-response effect on Postprandial glycemic control in insulin resistant individuals.plasma insulin concentration is measured over 6 hours by Randox clinical analyzer, analyzed with SAS mixed model.
Time Frame: 6 hour postprandial study over 4 periods
Population: study completer who finished all 4 treatments.
Measure: Mean (Standard Error); unit: microIU/mL
Arm/Group | Placebo | 10G STRB Powder | 20G STRB Powder | 40G STRB Powder
Number analyzed (Participants) | 21 | 21 | 21 | 21
microIU/mL | 63.9 (5.6) | 64.3 (5.6) | 60.2 (5.6) | 56.3 (5.6)

2. Secondary Outcome: Strawberry Dose-response Effect on Postprandial Oxidative Stress (Ox-LDL) in Insulin-resistant Men and Women in an Acute Postprandial Paradigm
Description: Postprandial plasma Ox-LDL concentration was measured by ELISA method. Normalizing responses to subjects own baseline (Time 0) was analyzed by SAS mixed model.
Time Frame: 6 hours postprandial study over 4 periods(treatments)
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Placebo | 10G STRB Powder | 20G STRB Powder | 40G STRB Powder
Number analyzed (Participants) | 21 | 21 | 21 | 21
U/L | -0.1 (0.8) | -0.3 (0.8) | -3 (0.8) | -0.17 (0.8)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Placebo | 10G STRB Powder | 20G STRB Powder | 40G STRB Powder
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
The study had the following limitations: the study was single blinded and lack of data on other non-anthocyanin strawberry polyphenols and their metabolites may yield additional insight on the relationship between strawberry polyphenols & bioactivity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No